CLINICAL TRIAL: NCT06122051
Title: Dynamic Chest X-ray With Simultaneous Spirometry
Acronym: DynaSSaur
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 322890; IRAS project ID: 322890 (Other: Health Research Authority)
Record Dates: First submitted 2023-10-19; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis
Keywords: Dynamic chest X-ray
MeSH Terms: conditions — Cystic Fibrosis | interventions — Spirometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP A: no significant underlying lung condition: No significant Underlying lung condition. An Asthma diagnosis requiring short-acting bronchodilators only will be eligible.
  For Dynamic Chest - x-ray and simultaneous Spirometry
  Interventions: Radiation: Dynamic chest x-ray; Diagnostic Test: Spirometry
- GROUP B: People with CF: Diagnosis of Cystic Fibrosis For Dynamic Chest x-ray and simultaneous spirometry. Retrospective review of Dynamic Chest-xray metrics and key clinical markers of CF as recorded by the annual review process
  Interventions: Radiation: Dynamic chest x-ray; Diagnostic Test: Spirometry

INTERVENTIONS:
Radiation: Dynamic chest x-ray — Group A and Group B- posterior-anterior dynamic chest x-ray film (Group A, This will represent an additional intervention not part of standard clinical care) (Group B, People with CF, already have this as part of their annual review process)
Diagnostic Test: Spirometry — Group A and Group B- Spirometry lung function test (Group A, This will represent an additional intervention not part of standard clinical care) (Group B, People with CF, already have this as part of their annual review process)

SUMMARY:
Dynamic chest X-ray (DCR) is a novel radiographic technique that enables us to visualise the movement of the chest and lungs in real-time by recording a series of x-ray images over 10-20 second interval. DCR provides an assessment of structures involved in respiration over a time period and could therefore provide us with insights into respiratory function. It may be possible that relating DCR to conventional breathing tests allows it to be used as a surrogate tool to measure lung function. Alternatively, it may provide different parameters of lung function which don't directly correlate with conventional testing, but are of themselves clinically relevant.

Cystic fibrosis (CF) is a genetic condition that results in the body producing thick , dehydrated secretions. It is usually characterised by a cycle of recurring lung infections and inflammation resulting in progressive lung damage. A key clinical investigation for people with cystic fibrosis (pwCF), and other chest conditions, is a spirometry breathing test. Despite spirometry's fundamental role in chest medicine it can be poorly tolerated.

In order to evaluate the utility of DCR as a tool for assessing lung function, it is important to be able to compare it to currently available pulmonary function tests such as spirometry. Previous studies have compared sequential lung function testing to DCR images; however, there may be significant variability in 2 separate manoeuvres as they are effort and technique dependent (i.e. when performing a DCR followed by spirometry or vice versa). Currently, there have been no studies that compare DCR with a simultaneous lung function test such as spirometry.

This observational, prospective, non-randomised, single centre , pilot study aims to address this issue by performing simultaneous spirometry and DCR to establish how DCR compares with spirometry in a healthy population of individuals. The investigators would seek to also perform the DCR with simultaneous spirometry in a cohort of pwCF, allowing for comparison between the two groups. Furthermore DCR imaging has been part of the annual review process for pwCF at Liverpool Heart and Chest Hospital since 2019. The study investigators therefore intend to review how changes in DCR metrics over time relate to changes in other key clinical markers of pwCF, such as spirometry. A questionnaire on patient experiences of DCR will be provided to study participants to be filled in after imaging acquisition.

DETAILED DESCRIPTION:
Dynamic chest X-ray (DCR) records images of the chest in motion in a 'recording' over 10-20 seconds. This is essentially a video x-ray of the chest and associated structures involved in breathing. The images acquired by the DCR can be processed using computer algorithm and key quantitative measures derived (such as diaphragm movement speed and changes in lung field area). Due to the way the X-ray is acquired, this is relatively lower radiation than other video caption imaging available (such as fluoroscopy). The time component of the imaging (vs static imaging) also opens up possibilities for clinical utilisation beyond imaging techniques that are already available without losing clinical information that a conventional static x-ray provides. The direct visualization of the chest and lung field in motion may therefore provide clinically relevant information about respiratory function. It may be possible that relating DCR to conventional lung function testing allows it to be used as a surrogate tool for assessing pulmonary function. Alternatively, it may provide different parameters of lung function that don't directly correlate with conventional testing but are of themselves clinically relevant.

Cystic fibrosis (CF) is an autosomal recessive genetic condition resulting in viscid, dehydrated luminal secretions. It has multi-system consequences but is usually characterised by a cycle of recurring lung infections and inflammation resulting in progressive lung damage. A key clinical investigation for people with cystic fibrosis (pwCF), as well as many other chest conditions, is a spirometry breathing test. Despite this spirometry can be poorly tolerated in individuals with underlying respiratory conditions. Patient factors combined with the ease and speed of acquiring DCR may mean it is better tolerated than conventional pulmonary function techniques such as spirometry. No previous studies have directly compared DCR with simultaneous breathing tests (such as spirometry). This is important as there can be significant variability in two different breathing manoeuvres such as used in breathing tests like spirometry. This means direct comparison is difficult when the tests are performed sequentially.

This study aims to address this by performing simultaneous spirometry and DCR to establish how DCR compares with spirometry in a healthy population of individuals. Study investigators also aim to perform DCR with simultaneous spirometry in a cohort of people with cystic fibrosis (pwCF), this would allow for comparison between the two groups. Furthermore the DCR has been part of Liverpool Heart and Chest Hospital's (LHCH) annual review process for pwCF since 2019. Study investigators therefore intend to review how changes in DCR metrics over time relate to other key clinical parameters for pwCF such as spirometry values. A questionnaire on patient experiences of DCR will be provided to patients after completion of the examinations, to be filled in at the time of investigation acquisition.

Principal research objective: to understand how DCR relates to a conventional assessment of lung function testing in the form of spirometry in both pwCF and those with no underlying lung health problems.

Secondary research objective: to understand how the relationship between metrics recorded by DCR imaging over time and key clinical markers of CF recorded in the annual review process, such as lung function recorded by spirometry.

Study design and methodology:

This observational, prospective, non-randomised, single centre , pilot study will be taking place at LHCH. The investigations will be performed in the DCR room of LHCH

Individuals will be asked to take part in the study if they (A) have no significant underlying lung condition or are (B) pwCF and are under the care of the LHCH CF team. The investigators are aiming to recruit 100 people in group (A) and 100 people in group (B). This study is exploratory work and is ultimately hypothesis generating and as such no formal statistical power calculation has been carried out. Target recruitment numbers are therefore based on a pragmatic assessment of the ability to recruit and measure successfully. LHCH has a cohort size of around 350 people with CF, of these 48 aren't attending locally. Approximately 22 will be excluded due to pregnancy or lung transplant. The projected DNA rate is around 30% and the projected exacerbation rate on attendance is about 20%. The projected cohort number therefore eligible for recruitment is around 157. In reality, this is a conservative estimate as those who do not attend annual review or who have an exacerbation usually then have a further face-to-face appointment arranged.

A poster campaign within the hospital will be used to recruit a healthy population with no underlying respiratory diagnosis. If interested they will contact the study team and be provided with a patient information sheet.

PwCF will be identified from LHCH hospital disease register and the CF coordinator will send out a letter to all pwCF inviting them to express interest in the study.

All participants will be encouraged to read the Patient information leaflet. Assessment of capacity to consent will be made by the consenting member of the investigating team who will be a General Medical Council registered physician, with up-to-date Good Clinical Practice and registered on the study delegation log. The same member will review the relevant inclusion and exclusion criteria to ensure recruitment is appropriate. If volunteers are happy to proceed a consent form will be filled in with the study team ensuring participants understand what is involved.

Advice from LHCH patient group (SURE group) has been sought in writing patient information sheets, consent forms, and the questionnaire. This is particularly relevant to group (A) where investigations involved in the study are in addition to standard care and to ensure participants fully understand what is involved.

Those individuals with no underlying lung condition will attend the radiology department at a pre-arranged slot to perform study investigations. PwCF attend face-to-face to complete an annual review once a year. Those consenting to be involved with the study will have the study investigations at this annual review attendance. At LHCH pwCF already have a DCR and Spirometry as part of routine clinical care therefore involvement with this study involves no further exposure to ionising radiation in the form of further X-rays.

Simultaneous DCR and spirometry acquisition:

Spirometry is a breathing test that involves blowing into a tube to work out the flow of air in the lungs; it is a safe examination, but some people may find the breathing exercises involved tiring. Participants will be seated on a stool for this test with their chest against the flat panel of the x-ray machine. In this position, they will be asked to hold a device with a tube to their mouth to blow into. A breathing test specialist will coach study participants through what is expected. For the actual blow tests instructions will be called out to perform the necessary manoeuvre (even if people have done them before). The test involves taking a deep breath in then blowing out as hard as possible into the tube until all air is expelled from their lungs. Study participants will have to perform at least 3 blows in total. The first 2 blow tests are spirometry only; If they and the investigating team are happy with the technique the investigators will progress to recording a simultaneous dynamic x-ray with the third blow attempt. This will be in exactly the same format, but the radiographer will press record whilst the breathing instructions are given. If participants need longer to perfect the technique of spirometry or have questions the study team will take longer to make sure that the participant is happy and the technique is good before recording the simultaneous x-ray. Each blow takes about 10-20 seconds and the x-ray will be recorded at the same time on the final blow.

After the investigations are performed the study participant will be asked to complete a short questionnaire in the radiology waiting room. The entire procedure including completing the questionnaire should take around 30 minutes.

The investigating team will record the x-ray and spirometry results as well as some basic information, such as age , sex, height and weight. This is the only participation required and individuals will not be asked to attend any further visits for the purposes of this study. The pwCF will also be consented for accessing medical records and investigations (to record key parameters of annual review including microbial colonisation, co-morbidities, and previous DCR metrics).

PwCF have been consulted by members of the investigating team to ensure that the study is designed to accommodate this group of individuals as best as possible. Individuals with no underlying health conditions have also been canvassed regarding their perspectives on the study.

Potential risks and burdens:

Exposure to ionising radiation carries the risk of developing malignancy. Detailed information on this, adhering to the guidance provided by the health research authority, has been included in the patient information Leaflet and reflected in the consent process. Dynamic chest radiography is CE-marked for thoracic imaging and is in routine clinical use as part of the annual review process for people with CF at LHCH. For pwCF this study carries no more exposure to ionising radiation than of routine clinical care.

DCR with simultaneous spirometry involves sitting in front of an X-ray plate whilst breathing in and out into the spirometer. This can cause occasional dizziness and or breathlessness. The procedure will be performed with the individual sitting on a stool with an accredited physiologist performing spirometry. Patients are screened against exclusion criteria prior to participation and are counselled by the physiologist as to the risks and potential side effects of spirometry.

Recruitment and informed consent:

Storage and personal data use during the study:

Whilst DCR data interpretation is carried out on workstations belonging to the manufacturer of the dynamic x-ray equipment, Konica Minolta, Inc., no personally identifiable data is stored on these workstations long-term and is deleted as per guidelines implemented by the radiology data manager at LHCH. The data will be transferred onto the workstation for analysis, and then deleted, in an automated process. Transfer is by the local Trust ethernet network.

Data is backed up on the local picture archiving and communication system (PACS) server and on a separate secure Trust server. Both of these are in keeping with local data storage policy. Case report forms will be kept within a locked cabinet, and stored in the Trust's Research Department, in accordance with standard operating procedures for the Trust. Electronic data will be stored on the local PACS server and on a local Trust server, both adhering to the Trust's data protection standards.

With the consent of patients (as per the consent form), quotations from the study questionnaire may be published.

No third-party persons outside the research team will have access to the study data. Study reference numbers will be used instead of personally identifiable information (such as names) in the documentation/databases.

Long-term arrangements for storage of data after the study has ended:

Anonymised data will be archived on a National Health Service computer, password protected and accessible only by members of the research team. Archived physical data will be stored within a locked cabinet in the Trust Research Department in accordance with local data governance standard operating procedure.

ELIGIBILITY:
Part A: Real-time paired DCR and Spirometry in Healthy cohort with no underlying respiratory diagnosis

Inclusion criteria:

* Age: ≥ 17 years old and <_ 50 years old
* No underlying respiratory illness (chronic or acute). Individuals with an Asthma diagnosis requiring short-acting bronchodilators only will be eligible
* Able to provide informed consent

Exclusion criteria:

General exclusion criteria:

Any of:

* Potentially pregnant or lactating
* Inability to provide informed consent
* Unable or unwilling to sit to perform Dynamic chest x-ray/Spirometry in the radiology department
* Unable or unwilling to follow Spirometry breathing instructions (e.g., holding breath or taking a deep breath)
* Unable to perform reproducible spirometry and/or full pulmonary function studies within American Thoracic Society and European Society joint criteria
* Significant radiation exposure within the last year (for example, numerous CT scans of chest)
* Involved, either currently or recently, in other studies involved non-routine exposure to sources of ionising radiation
* Any serious or active medical or psychiatric illness, which in the opinion of the investigators, would interfere with subject treatment, assessment, or compliance with the protocol
* Inability to complete spirometry in 20 seconds.
* Current Chest infection

Spirometry exclusion criteria

Any of:

* Unstable cardiovascular status, recent myocardial infarction or pulmonary embolism (within 6 weeks)
* Haemoptysis of unknown aetiology (within 6 weeks)
* Pneumothorax (present, or occurring within 6 weeks)
* Within 24 hours of bronchoscopy
* Thoracic, abdominal or cerebral aneurysm
* Recent eye surgery or increased intraocular pressure
* Recent thoracic or abdominal surgery
* Acute nausea, vomiting or diarrhoea
* Pregnancy
* Undergoing treatment for tuberculosis

Part B: Real-time paired DCR and spirometry in a CF subgroup

Inclusion criteria:

* Age: ≥ 17 years old and
* Attending the adult CF Unit at Liverpool heart and Chest Hospital and
* Confirmed CF diagnosis (positive sweat test in childhood and by genotyping) and
* Able to provide informed consent

General exclusion criteria, same as Group A (see above) plus:

* Recipient of Lung transplant
* Current exacerbation Spirometry exclusion criteria (same as for Group A, see above)

Ages: 17 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Individuals will be asked to take part in the study if they (A) have no significant underlying lung condition or (B) have cystic fibrosis and are under the care of the Liverpool Heart and Chest Hospital team
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Correlation between Dynamic chest X-ray (DCR) metrics And Spirometry metrics in people with Cystic fibrosis and those with no underlying respiratory conditions | During the test (simultaneous acquisition of dynamic chest X-ray and Spirometry)
  DCR metrics as calculated by software analysis of DCR imaging. This includes: projected lung area, diaphragm movement and signal density of the image. Spirometry metrics: e.g forced expiratory volume at one second (FEV1) and forced vital capacity (FVC)

SECONDARY OUTCOMES:
Correlation between DCR metrics and Spirometry metrics over time, as recorded in annual review CF clinic attendance (non-simultaneous) | Day of annual review attendance up to 48 months prior (first DCR acquisition 2019)
  Patients with CF attend an annual review clinic once a year. This review includes a DCR and spirometry. The DCR metrics data is produced through software analysis of original DCR images and includes: projected lung area, diaphragm movement and signal density of the image. At this annual review people with CF also have spirometry. Spirometry metrics: e.g FEV1 and FVC.

OTHER OUTCOMES:
Correlation between DCR metrics and BMI for people with CF | Day of annual review clinic attendance and up 48 months prior (first DCR acquisition 2019)
  Patients with CF attend an annual review clinic once a year. This review includes a DCR as well as the record of other key clinical markers of CF. DCR metrics are produced through software analysis of original DCR images and include: projected lung area and diaphragm movement as well as signal density. From the annual review clinic attendance key CF data is recorded including BMI
Correlation between DCR metrics and microbial colonisation for people with CF | Day of annual review clinic attendance and up 48 months prior (first DCR acquisition 2019)
  Patients with CF attend an annual review clinic once a year. This review includes a DCR as well as the record of other key clinical markers of CF. DCR metrics are produced through software analysis of original DCR images and include: projected lung area and diaphragm movement as well as signal density. From the annual review clinic attendance key CF data is recorded including microbial colonisation
Correlation between DCR metrics and co-morbidities for people with CF | Day of annual review clinic attendance and up 48 months prior (first DCR acquisition 2019)
  Patients with CF attend an annual review clinic once a year. This review includes a DCR as well as the record of other key clinical markers of CF. DCR metrics are produced through software analysis of original DCR images and include: projected lung area and diaphragm movement as well as signal density. From the annual review clinic attendance key CF data is recorded including CF comorbidities
Correlation between DCR metrics and key CF respiratory medication for people with CF | Day of annual review clinic attendance and up 48 months prior (first DCR acquisition 2019)
  Patients with CF attend an annual review clinic once a year. This review includes a DCR as well as the record of other key clinical markers of CF. DCR metrics are produced through software analysis of original DCR images and include projected lung area and diaphragm movement as well as signal density. From the annual review clinic attendance key CF respiratory medication date to include Nebulised therapy, modulator therapy, steroids, mucolytics, inhalers

CONTACTS AND LOCATIONS:
Overall Officials: David AP Green, MbChb, Principal Investigator — David Green

IPD SHARING:
Plan to Share IPD: No
No There is no plan to make data widely available. However, should a legitimate request be made by researchers with data protection legislation equivalent to United Kingdom General Data Protection Regulations (GDPR), this would be considered. Governance procedures to anonymise all identifiable details would be required for individual participant data, but protocols etc would be shared after the publication of the study.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT06122051/Prot_SAP_000.pdf
  • Informed Consent Form: People with CF (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT06122051/ICF_001.pdf
  • Informed Consent Form: Control group (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT06122051/ICF_002.pdf